CLINICAL TRIAL: NCT05581667
Title: The Immediate Effects of Post Isometric Relaxation Techniques In Hospital Employees With Neck Pain: A Randomised Control Trial
Brief Title: The Immediate Effects of Post Isometric Relaxation Techniques
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bulent Ecevit University (Other)
Responsible Party: Principal Investigator, Sanem ŞENER, Principal Investigator, Bulent Ecevit University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Immediate PIR
Record Dates: First submitted 2022-10-12; First posted 2022-10-14 (Actual); Last update posted 2023-12-28 (Actual); Status verified 2023-12

CONDITIONS: Neck Pain
Keywords: neck pain; Post isometric relaxation; hospital employees; pain threshold
MeSH Terms: conditions — Neck Pain

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- PIR Group (Experimental): PIR Group participants will be given a one-time PIR Technique for each of the neck and upper back muscles, right after the classical Swedish massage is applied to the cervical region and upper back area.
  Interventions: Other: post isometric relaxation; Other: Swedish Massage
- Control Group (Experimental): Control group participants will receive classical Swedish massage only to the cervical and upper thoracic region.
  Interventions: Other: Swedish Massage

INTERVENTIONS:
Other: post isometric relaxation — PIR is performed by first passively lengthening the muscle, then having the patient lightly contract (10-20% of maximum) against resistance for 5 seconds passively before exhaling and relaxing the muscle and repeated. The clinician then takes up the slack within the muscle and repeats the technique 3 to 5 times
  Arms: PIR Group
Other: Swedish Massage — classic Swedish massage for the cervical and upper thoracic region. Massage is a method that is applied to superficial soft tissues such as muscles, skin, ligaments and fascia and structures located under the superficial tissues and aims to relax.

SUMMARY:
Aim: The aim of this study is to investigate the immediate effects of Post Isometric Relaxation (PIR) Technique on pain threshold, pain severity and joint range of motion of the cervical region in healthcare workers with neck pain.

Method: A total of 30 male and female participants aged 20-45 were randomly divided into two groups (Post Isometric Relaxation (PIR) Technique and Control Group). PIR group participants were under a single session of PIR application with 10 repetitions to m.supraspinatus, the upper part of the m.trapeze and m.levator scapula in addition to classical Swedish massage for neck and upper thoraric region. Control group participants received only classical Swedish massage to the cervical and upper thoracic region. Pain severity (Visual Analog Scale), Pain threshold (digital algometer), range of servical motion (goniometer) were measured at baseline and immediately after the single-session PIR Techniques.

DETAILED DESCRIPTION:
Neck pain is the second most common musculoskeletal problem in the world after low back pain in terms of disability and health expenditures. Occupational groups with the highest incidence of neck pain include those working in a hospital environment, office workers, and manual workers.

Post Isometric Relaxation Technique (PIR) is a Muscle Energy Technique (MET) and is used by physiotherapists to relax muscles, reduce pain and increase range of motion. The PIR Technique provides its neurological effects through autogenic inhibition, which results in relaxation in the agonist muscle by inhibiting contraction with the stimuli sent by the group Ib fibers originating from the Golgi tendon organ of the agonist muscle to the medulla spinalis during static stretching.

The aim of our study is to investigate the instantaneous effect of PIR Technique on pain threshold, pain intensity and joint range of motion (neck flexion, extension, right and left rotation, right and left lateral flexion) in hospital workers with neck pain.

This experimental study, which was planned as randomized and single-blind, was planned to be carried out with a total of 30 volunteer participants, male and female, working in a private hospital in Istanbul between 7 October 2022 and 10 December 2022.

ELIGIBILITY:
Inclusion Criteria:

* be a hospital worker
* complaining of neck pain for at least 3 months
* pain intensity at rest is 4 out of 10 according to VAS assessment
* volunteer to participate in the study

Exclusion Criteria:

* Having neck pain after trauma to the neck in the last 6 months
* presence of neurological signs; neck pain that has spread to the arm and fingers
* have had spinal surgery
* shoulder pathology

Ages: 20 Years to 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2022-10-07 (Actual); Primary Completion 2022-11-07 (Actual); Study Completion 2022-12-10 (Actual)

PRIMARY OUTCOMES:
Pain threshold assessment | 30 min
  Digital algometer (JTECH Commander ™ Algometer with 0.5 cm2 tip) device was used. After training by showing the measuring instrument to the participants, pressure will be applied to a place outside the assessment area to introduce the feeling of pressure. He will be told to give a "stop" command as soon as the pain is first felt. This process will be applied 3 times to ensure that the participants adapt to the pressure to be applied during the evaluation. Before and immediately after the applications, all participants felt the pain for the first time with a speed of 10 N/s over the sensitive points of the m.trapezius pars descendes, m.levator Scapula, m.Rrhomboideus Major, M.Sternocleidomasteideus, suboccipital region, M. Infraspinatus, M. Multifidius muscles. will be increased so far. The measurement was terminated with the "Stop" command and a total of 3 measurements will be made and the average value seen on the screen will be recorded.
Pain severity assessment | 30 min
  After explaining that '0 is no pain, 10 is the most severe pain', all participants will be asked to mark the intensity of pain they feel on the 10 cm horizontal Visual Analog Scale (VAS) before and immediately after the application.
Joint Range of Motion | 30 min
  In order to evaluate the range of motion of the cervical vertebrae, measurements will be made before and immediately after the applications using a universal goniometer and according to Kendall-Mc Creary criteria. The fixed arm, pivot point and movable arm of the goniometer will be placed in certain reference areas in the measurement that starts when the participant is in a sitting position. Measurements of cervical flexion, extension, right and left lateral flexion, right and left rotation will be recorded after the participant's active movements, the angle value at the end of the movement, the active joint range of motion measurement.

CONTACTS AND LOCATIONS:
Locations (1):
- Zonguldak Bülent Ecevit University, Zonguldak, Kozlu, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cohen SP. Epidemiology, diagnosis, and treatment of neck pain. Mayo Clin Proc. 2015 Feb;90(2):284-99. doi: 10.1016/j.mayocp.2014.09.008. PMID 25659245
- [Background] Page P. Cervicogenic headaches: an evidence-led approach to clinical management. Int J Sports Phys Ther. 2011 Sep;6(3):254-66. PMID 22034615